CLINICAL TRIAL: NCT04157283
Title: Sexual Dysfunction in Patients With Relapsing Remitting Multiple Sclerosis and Associated Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 3
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis; Sexual Dysfunction
MeSH Terms: conditions — Multiple Sclerosis; Sexual Dysfunction, Physiological | interventions — Evoked Potentials, Visual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 60 male patients
  Interventions: Diagnostic Test: MRI brain, visual evoked potential, Cerebrospinal Fluid, Sexual dysfunction measure, Depressive symptoms assessment and Multiple Sclerosis Quality of Life-54(MSQOL-54)
- Group 2: 60 female patients
  Interventions: Diagnostic Test: MRI brain, visual evoked potential, Cerebrospinal Fluid, Sexual dysfunction measure, Depressive symptoms assessment and Multiple Sclerosis Quality of Life-54(MSQOL-54)

INTERVENTIONS:
Diagnostic Test: MRI brain, visual evoked potential, Cerebrospinal Fluid, Sexual dysfunction measure, Depressive symptoms assessment and Multiple Sclerosis Quality of Life-54(MSQOL-54) — 1. Neurophysiological Evaluation:
     Visual Evoked Potential (VEP).
  2. Imaging Evaluation:
     Conventional MRI.
  3. Cerebrospinal Fluid (CSF):
  4. Sexual dysfunction measure: through the international index of erectile function (IIEF), female sexual function questionnaire (SFQ) and the sexual Quality of life male and female version (SQoL) (American Psychiatric Association, 1994).
  5. Depressive symptoms assessment through The BDI (The Beck Depression Inventory) which is the most common instrument measuring the severity of depression.
  6. Fatigue symptoms were evaluated through fatigue subscale of Multiple Sclerosis Quality of Life-54(MSQOL-54).

SUMMARY:
This work aims to:

1. Investigate and correlate Sexual Dysfunction in relapsing-remitting Multiple Sclerosis patients with specific focus on

   1. Specific neurologic deficit.
   2. Depressive symptoms.
   3. Comorbid factors.
   4. Fatigue symptoms.
2. To investigate the impact of Sexual dysfunction on Sexual Quality of Life (SQoL).
3. To search for possible gender difference.

DETAILED DESCRIPTION:
The present study is a cross sectional study on 120 MS adolescent patients meeting the McDonald's criteria; 60 male cases and 60 female cases recruited from Mansoura University Hospitals, Egypt.

All patients were subjected to the following:

1. Clinical Evaluation:

   1. Thorough neurological examination.
   2. Cognitive functions by Minimental State Examination (MMSE).

   e. Expanded Disability Severity Scale (EDSS).
2. Neurophysiological Evaluation:

   a. Visual Evoked Potential (VEP).
3. Imaging Evaluation:

   a. Conventional MRI.
4. Cerebrospinal Fluid (CSF):
5. Sexual dysfunction measure: through the international index of erectile function (IIEF), female sexual function questionnaire (SFQ) and the sexual Quality of life male and female version (SQoL) (American Psychiatric Association, 1994).
6. Depressive symptoms assessment through The BDI (The Beck Depression Inventory) which is the most common instrument measuring the severity of depression.
7. Fatigue symptoms were evaluated through fatigue subscale of Multiple Sclerosis Quality of Life-54(MSQOL-54).

ELIGIBILITY:
Inclusion Criteria:

* 120 MS adolescent patients meeting the McDonald's criteria; 60 male cases and 60 female cases recruited from Mansoura University Hospitals

Exclusion Criteria:

The exclusion criteria:

* Active relapse or relapse during 30 day prior to survey due to significant changes in all life activities during this period including sexuality.
* EDSS score equal or higher than 6.5.
* Current pregnancy in female patients.
* Form of the disease other than RRMS.
* Patients with any sort of cognitive impairment preventing them from understanding Questionnaire.
* Poorly controlled concomitant diseases were excluded.
* Patients with past history of any sexual problems prior to the first MS attack.
* UN married Patients.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 120 MS adolescent patients meeting the McDonald's criteria; 60 male cases and 60 female cases
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The Sexual Quality of Life-Male (SQOL-M) | 24-48 hours
  Assesses the relationship between male sexual dysfunction and quality of life. It contains 11 items, each items are scored from 1 to 6 points (worst to best)-completely Agree = 1 to Completely Disagree = 6. The total score can range from 11 to 66 points.
The Sexual Quality of Life-Female (SQOL-F) | 24-48 hours
  Assesses the relationship between female sexual dysfunction and quality of life. It consists of 18 items, rated using a six-point scale (completely agree to completely disagree). The total score can range from 18 to 108 points. Higher scores indicate better female sexual quality of life.
The international index of erectile function (IIEF) | 24-48 hours
  It's formed of 15 questions about main domains of male sexual function and each one had a score of 0-5 but used in Arabic translation.

SECONDARY OUTCOMES:
Beck's Depression Inventory | 24-48 hours
  The highest possible total for the whole test would be sixty-three. The lowest possible score for each question is zero, the lowest possible score for the test would be zero. This would mean you circles zero on each question. You can evaluate your depression according to the score below:
  1-10 score considered normal. 11-16 score considered Mild depression. 17-20 score considered borderline clinical depression. 21-30 score considered moderate depression. 31-40score considered severe depression. Over 40 score considered extreme depression
Fatigue symptoms | 24-48 hours
  Modified Fatigue Impact Scale (MFIS):
  Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities. The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales but used in Arabic translation.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Result] 2) Chan,K.,& Tsang, L. (2011). Promote healthy eating among adolescents:A Hong Kong study . Journal of Consumer Marketing, 28(5), 354-362.
- [Result] Fangerau T, Schimrigk S, Haupts M, Kaeder M, Ahle G, Brune N, Klinkenberg K, Kotterba S, Mohring M, Sindern E; Multiple Sclerosis Study Group. Diagnosis of multiple sclerosis: comparison of the Poser criteria and the new McDonald criteria. Acta Neurol Scand. 2004 Jun;109(6):385-9. doi: 10.1111/j.1600-0404.2004.00246.x. PMID 15147460
- [Result] Fraser C, Mahoney J, McGurl J. Correlates of sexual dysfunction in men and women with multiple sclerosis. J Neurosci Nurs. 2008 Oct;40(5):312-7. doi: 10.1097/01376517-200810000-00010. PMID 18856253
- [Result] Freedman MS, Thompson EJ, Deisenhammer F, Giovannoni G, Grimsley G, Keir G, Ohman S, Racke MK, Sharief M, Sindic CJ, Sellebjerg F, Tourtellotte WW. Recommended standard of cerebrospinal fluid analysis in the diagnosis of multiple sclerosis: a consensus statement. Arch Neurol. 2005 Jun;62(6):865-70. doi: 10.1001/archneur.62.6.865. PMID 15956157
- [Result] Kesselring J, Beer S. Symptomatic therapy and neurorehabilitation in multiple sclerosis. Lancet Neurol. 2005 Oct;4(10):643-52. doi: 10.1016/S1474-4422(05)70193-9. PMID 16168933
- [Result] Lew-Starowicz M, Gianotten WL. Sexual dysfunction in patients with multiple sclerosis. Handb Clin Neurol. 2015;130:357-70. doi: 10.1016/B978-0-444-63247-0.00020-1. PMID 26003254
- [Result] Marrie RA. Environmental risk factors in multiple sclerosis aetiology. Lancet Neurol. 2004 Dec;3(12):709-18. doi: 10.1016/S1474-4422(04)00933-0. PMID 15556803
- [Result] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Result] Zivadinov R, Zorzon M, Bosco A, Bragadin LM, Moretti R, Bonfigli L, Iona LG, Cazzato G. Sexual dysfunction in multiple sclerosis: II. Correlation analysis. Mult Scler. 1999 Dec;5(6):428-31. doi: 10.1177/135245859900500i610. PMID 10618700